CLINICAL TRIAL: NCT02481427
Title: Total Knee Arthroplasty Versus Unicondylar Knee Arthroplasty: a Randomized, Double-blind Multicenter Trial
Brief Title: Finnish Unicompartmental and Total Knee Arthroplasty Investigation
Acronym: FUNCTION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Jani Knifsund, MD, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T127/2015
Record Dates: First submitted 2015-06-15; First posted 2015-06-25 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Total; Unicondylar; Osteoarthritis; Arthroplasty; Replacement; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Knee Replacement (Experimental): TKA is performed through a standard medial parapatellar incision, which provides easy access to the knee joint. Skin incision is done to midline. Intramedullary guide is used for alignment of femoral and tibia saw cuts and component positions. Components will be cemented in position. The patella will not be resurfaced. Intraoperative local infiltration analgesia (LIA) is used for postoperative pain management. Drain is not used.
  Interventions: Procedure: Total Knee Replacement
- Unicondylar Knee Replacement (Experimental): UKA involves only the replacement of affected medial compartment. In the study, the operation will be performed through standard medial parapatellar incision with midline skin incision, but the knee joint and fascia will be opened like in standard Oxford minimally invasive incision. The procedure will be performed by using Oxford Microplasty instrumentation and following Microplasty surgical technique (Biomet Orthopedics). Intraoperative local infiltration analgesia is used for postoperative pain management. Drain is not used.
  Interventions: Procedure: Unicondylar Knee Replacement

INTERVENTIONS:
Procedure: Unicondylar Knee Replacement — UKA involves only the replacement of affected medial compartment. In the study, the operation will be performed through standard medial parapatellar incision with midline skin incision, but the knee joint and fascia will be opened like in standard Oxford minimally invasive incision. The procedure will be performed by using Oxford Microplasty instrumentation and following Microplasty surgical technique (Biomet Orthopedics). Intraoperative local infiltration analgesia is used for postoperative pain management. Drain is not used.
  Other Names: Oxford phase 3, unicondylar knee artrhoplasty
  Arms: Unicondylar Knee Replacement
Procedure: Total Knee Replacement — TKA is performed through a standard medial parapatellar incision, which provides easy access to the knee joint. Skin incision is done to midline. Intramedullary guide is used for alignment of femoral and tibia saw cuts and component positions. Components will be cemented in position. The patella will not be resurfaced. Intraoperative local infiltration analgesia (LIA) is used for postoperative pain management. Drain is not used.
  Other Names: Triathlon CR
  Arms: Total Knee Replacement

SUMMARY:
Unicondylar knee arthroplasty (UKA) can be used as the treatment of knee OA isolated to a single compartment instead of TKA. Both UKA and TKA have been used for decades as a treatment of knee OA. However, operative indications for TKA and UKA overlaps, but they are not similar. Therefore, the outcome or survivorship of these procedures cannot be compared directly.

Some advantages of UKA over TKA have been reported, including faster recovery time, reduced perioperative morbidity and mortality, a subjective preference of feeling more normal knee, lower cost and improved return to work and sport. On the other side national arthroplasty registers consistently report around a threefold increase in crude cumulative revision rate at 8 to 10 years for UKA compared with TKA 7-10.

The aim of this study is to compare functional, clinical, patient satisfaction, and implant survival results of cementless UKA with those of cemented TKA at 2 months, 1, 2, 5 and 10 years after the procedure. The study design is a multicenter, double-blind and randomized trial of knee replacement patients. The primary outcome is the Oxford Knee Score (OKS) and Knee Injury and Osteoarthritis Outcome Score (KOOS) at 2 year.

DETAILED DESCRIPTION:
Background Knee osteoarthritis (OA) is a common joint disease, which may cause severe pain and lead to a reduced quality of life. It has been shown that the prevalence of symptomatic OA in those aged 60 and above was 9.6% in men and 18% in women. Primary treatment of knee OA is conservative including physical activity, exercise and analgesics. Meta-analysis shows small to moderately sized effects of exercise on pain and function. Total knee arthroplasty (TKA) is the gold standard option for the treatment of painful OA of the knee when conservative treatment is not sufficient.

Unicondylar knee arthroplasty (UKA) can be used as the treatment of knee OA isolated to a single compartment instead of TKA. Both UKA and TKA have been used for decades as a treatment of knee OA. However, operative indications for TKA and UKA overlaps, but they are not similar. Therefore, the outcome or survivorship of these procedures cannot be compared directly.

Some advantages of UKA over TKA have been reported, including faster recovery time, reduced perioperative morbidity and mortality, a subjective preference of feeling more normal knee, lower cost and improved return to work and sport. On the other side national arthroplasty registers like the National Joint Registry of England and Wales (NJR), the Australian Orthopaedic Association National Joint Replacement Registry (AOANJRR), the Swedish Knee Arthroplasty Register (SKAR), and the Finnish Arthroplasty Register (FAR) consistently report around a threefold increase in crude cumulative revision rate at 8 to 10 years for UKA compared with TKA 7-10. Few reports have been published about patient-perceived outcomes following TKA compared with UKA. Newman et all compared fixed bearing UKA to TKA and published better range of movement (ROM) after UKA. Sun PF et all compared mobile bearing UKA to fixed bearing TKA. They didn't had significant difference in ROM or Knee Society score (KSS) postoperatively after mean 52 months follow-up, but in TKA group had significantly more postoperative deep vein thrombosis and more blood loss.

A study comparing cemented UKA (Oxford, Biomet) and TKA, have been published using patient-perceived outcome measures, but the study protocol lacks of blinding. There is no published randomized controlled, double-blind trial which compares patient-perceived outcomes after TKA and UKA.

Oxford mobile bearing UKA is most used unicondylar prosthesis according to national registries. The most common reason for revision of UKA according to NJR is aseptic loosening, accounting for up to 48% of all UKA revisions. Other reasons for UKA revision in Finland where malalignment, prosthesis fracture, instability, infection, fracture, patella complication and other reasons (35%). A randomized controlled trial of 62 knees comparing cemented and cementless Oxford UKA has demonstrated a greatly reduced incidence of tibial radiolucencies with similar functional outcomes at 1 year 15. Cementless Oxford unicondylar knee is relative new product and was developed to address problems related to cement fixation, and has been demonstrated in a randomised study to have similar clinical outcomes with fewer radiolucencies than observed with the cemented device. New Zealand Joint Registry (NZJR) data shows revision rate 1,37/100 component years for cemented Oxford phase 3 and 0,72/100 component years for cementless Oxford phase 3 UKA. The uncemented Oxford UKA has a significantly lower revision rate than the overall mean of 1.27 /100 observer component years. Also the NJR show better survivorship for cementless unicondylar arthroplasty compared to cemented unicondylar arthroplasty. On the other hand cementless TKA shows lower survivorship compared cemented TKA in Finnish Arthroplasty Register (FAR). There are no published randomized controlled, double-blind trial which compare patient-perceived outcomes after cemented TKA and cementless Oxford UKA.

The aim of the study The aim of this study is to compare functional, clinical, patient satisfaction, and implant survival results of cementless UKA with those of cemented TKA at 2 months, 1, 2, 5 and 10 years after the procedure.

Study setting The study design is a multicenter, double-blind and randomized trial of knee replacement patients. Arthroplasty procedures will be performed by experienced knee surgeons who are experienced in both UKA and TKA operations. As UKA we will use cementless Oxford phase 3 mobile bearing prosthesis with Microplasty instrumentation (Biomet) and as TKA cemented Triathlon CR condylar prothesis (Stryker). According to power analysis, we are going to recruit 140 patients from 3 orthopedic units in Finland. Participants will be randomized to UKR or TKR.

Study participants Participants with anteromedial osteoarthritis of knee will be included in the study. Patients must be applicable for both a medial UKR and TKR.

Recruitment and consent Potential patients will be contacted in outpatient clinics by the participating orthopedic surgeon. At this stage patients will be provided with an 'Invitation letter' and a information sheet which will explain why they have been approached and will provide further details about the study. Those patients, who voluntary will take part to the study, will be screened for inclusion and exclusion criteria. If the patient is appropriate for the study, pre-assessment clinic appointment will be organized. The pre-assessment appointments are routine appointment for a short time before their scheduled operation date.

Study assessments Preoperative assessments will include a patient reported questionnaire examining pain, other Symptoms, function in daily living, function in sport and recreation and knee related Quality of life. (OKS and KOOS). Also a clinical assessment of range of motion and function of the knee, will be carried out. Preoperative weight bearing X-rays knees 20 degrease flexion, valgus stress x-rays and mechanical axis will also be taken.

After the operation, the operative details will be recorded and routine postoperative radiographs collected. Operative details will be sealed and saved. Code will be opened and randomization will be cancelled only if it's necessary. Reasons which might result in cancellation of randomization are, for example, symptoms of the operated knee which might require revision arthroplasty. Cancellation of randomization occurs also if the patient wants to discontinue participating to the study.

Control outpatient policlinic appointment will be arranged for the clinical examination at 2 months, 1, 2, 5 and 10 years post operation. Outpatient controls will be carried out by orthopedic surgeons, who are not aware which type of operation -UKA or TKA - was performed. Range of movement and stability are assessed. The radiographs are not available for the patient at the outpatient policlinic, but they are controlled by radiologists and the orthopedic surgeon to complications. Patients are informed of any surgical complications or possible abnormal findings in X-rays, and are treated using standard methods.

A postal questionnaire (containing the 15D, OKS and KOOS) will be sent out at 2 months, 1, 2, 5 and 10 years post randomization. Additional clinical appointments (if needed) will be performed by surgeon not participating study operations or controls.

Randomisation

2 to 24 hours before the operation, if a patient is confirmed to be eligible for the trial, the surgeon opens an envelope containing the study-group assignment (TKA or UKA). The assignment will not be revealed to the patient. The sequentially numbered, sealed envelopes will prepared by a statistician with no involvement in the clinical care of patients in the trial. Randomizations will be performed in a 1:1 ratio with a block size of 4. The randomization sequence involved stratification according to age (45 to 60 or 61 to 79 years of age), sex, and preoperative OKS (0-17, 18-27, or 28-48). Only the orthopedic surgeon and other staff in the operating room will be aware of the group assignment, and they do not participate in further treatment or follow-up of the patient.

Total knee replacement procedure TKA is performed through a standard medial parapatellar incision, which provides easy access to the knee joint. Skin incision is done to midline. Intramedullary guide is used for alignment of femoral and tibia saw cuts and component positions. Components will be cemented in position. The patella will not be resurfaced. Intraoperative local infiltration analgesia (LIA) is used for postoperative pain management. Drain is not used.

Partial knee replacement procedure UKA involves only the replacement of affected medial compartment. In the study, the operation will be performed through standard medial parapatellar incision with midline skin incision, but the knee joint and fascia will be opened like in standard Oxford minimally invasive incision. The procedure will be performed by using Oxford Microplasty instrumentation and following Microplasty surgical technique (Biomet Orthopedics). Intraoperative local infiltration analgesia is used for postoperative pain management. Drain is not used.

Safety The study participants have symptomatic medial knee OA and have failed conservative treatment. Patients, which are suitable for knee replacement have been selected from outpatient clinic. The operation will be performed as standard knee replacement.

The study participants will be informed of the risks associated with anesthesia and knee replacement surgery. Potential intra- or perioperative complication are; anesthesia-related complications, wound infection, bleeding, fracture, rupture of collateral or patellar ligament, thrombo-embolic complications, death, ongoing pain, and deterioration of existing co-morbidity.

Surgical long-term complications following the knee replacement are loosening of implant, lack of osteointegration of a cementless implant, periprosthetic fracture, luxation- or wear of bearing, infection, adverse knee pain 12 months after operation, knee stiffness, and lateral compartment OA in UKA. These complications may need surgery as revision, open debridement, washout or as worse even amputation.

Ethics and study registration We have approval of the institutional review board of Ethics Committee, Hospital District of Southwest Finland.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic medial knee OA with exposed bone on both femur and tibia.
* Age 45 to 79.
* Failed conservative treatment of knee OA.
* Mechanical axis 5 to 15 degrees varus.
* Functionally intact anterior cruciate ligament.
* Full thickness lateral cartilage present
* Correctable intra-articular varus deformity in knee 20 degrees flexion
* American Society of Anesthesiologists Physical Status Classification System (ASA) of 1, 2 or 3.

Exclusion Criteria:

* Rheumatoid arthritis or, other inflammatory disorders.
* Osteonecrosis
* Osteochondritis dissecans
* Symptomatic hip or spinal pathology
* Previous knee surgery other than diagnostic arthroscopy and medial menisectomy
* Previously had infectious arthritis
* Have significant damage to the patella-femoral joint especially on the lateral facet, patellar subluxation or concave patella.
* Previous ligament injury and instability
* Range of movement not within 15-100 degrees.
* Patient is planned to undergo simultaneous bilateral knee arthroplasty.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 2 months to 10 years
  Questionnaires will be collected also at 2 months, 1 year, 2 year, 5 and 10 years. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). KOOS is responsive to change following non-surgical and surgical interventions 17.
Oxford Knee Score (OKS) | 2 months to 10 years

SECONDARY OUTCOMES:
15D | 2 months to 10 years
  The health-related quality of life (HRQoL) instrument.
Knee Society Score (KSS) | 2 months to 10 years
  Range of Motion and Function
Radiographic features including signs of potential failures, including loosening and periprosthetic fracture | 2 months to 10 years
complications | 2 months to 10 years
  Anesthesia-related complications, wound infection, bleeding, fracture, rupture of collateral or patellar ligament, thrombo-embolic complications, death, ongoing pain, and deterioration of existing co-morbidity. According to Clavien-Dindo Classification of Surgical Complications
revision rate | 2 months to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Tuukka Niinimäki, MD PhD, Principal Investigator — Oulu University Hospital; Heikki Nurmi, MD, Principal Investigator — Central Finland Central Hospital; Alar Toom, MD PhD, Principal Investigator — Central Finland Central Hospital; Jani Knifsund, MD, Principal Investigator — Turku University Hospital; Keijo Mäkelä, Adj. Prof., Study Director — Turku University Hospital
Locations (3):
- Finland (3):
  - Central Finland Central Hospital, Jyväskylä
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku

REFERENCES:
- [Background] Bedson J, Jordan K, Croft P. The prevalence and history of knee osteoarthritis in general practice: a case-control study. Fam Pract. 2005 Feb;22(1):103-8. doi: 10.1093/fampra/cmh700. Epub 2005 Jan 7. PMID 15640302
- [Background] Fransen M, McConnell S. Land-based exercise for osteoarthritis of the knee: a metaanalysis of randomized controlled trials. J Rheumatol. 2009 Jun;36(6):1109-17. doi: 10.3899/jrheum.090058. Epub 2009 May 15. PMID 19447940
- [Background] Zipple J, Meyer-Ralfs M. Themistocles Gluck (1853-1942), pioneer in endoprosthetics. Z Orthop Ihre Grenzgeb. 1975 Feb;113(1):134-9. PMID 1098295
- [Background] Insall J, Walker P. Unicondylar knee replacement. Clin Orthop Relat Res. 1976 Oct;(120):83-5. PMID 975670
- [Background] Lombardi AV Jr, Berend KR, Walter CA, Aziz-Jacobo J, Cheney NA. Is recovery faster for mobile-bearing unicompartmental than total knee arthroplasty? Clin Orthop Relat Res. 2009 Jun;467(6):1450-7. doi: 10.1007/s11999-009-0731-z. Epub 2009 Feb 19. PMID 19225852
- [Background] Brown NM, Sheth NP, Davis K, Berend ME, Lombardi AV, Berend KR, Della Valle CJ. Total knee arthroplasty has higher postoperative morbidity than unicompartmental knee arthroplasty: a multicenter analysis. J Arthroplasty. 2012 Sep;27(8 Suppl):86-90. doi: 10.1016/j.arth.2012.03.022. Epub 2012 May 4. PMID 22560653
- [Background] Niinimaki T, Eskelinen A, Makela K, Ohtonen P, Puhto AP, Remes V. Unicompartmental knee arthroplasty survivorship is lower than TKA survivorship: a 27-year Finnish registry study. Clin Orthop Relat Res. 2014 May;472(5):1496-501. doi: 10.1007/s11999-013-3347-2. Epub 2013 Nov 19. PMID 24249531
- [Background] NJR. National Joint Registry for EnglandWales and Northern Ireland 10th annual report, 2013. 2013;10.
- [Background] SKAR. The Swedish Knee Arthroplasty Register Annual Report. 2012. 2012.
- [Background] AOANJRR. Australian Orthopaedic Association National Joint Replacement Registry Annual Report. 2011. 2011.
- [Background] Sun PF, Jia YH. Mobile bearing UKA compared to fixed bearing TKA: a randomized prospective study. Knee. 2012 Mar;19(2):103-6. doi: 10.1016/j.knee.2011.01.006. Epub 2011 Feb 22. PMID 21345681
- [Background] Newman JH, Ackroyd CE, Shah NA. Unicompartmental or total knee replacement? Five-year results of a prospective, randomised trial of 102 osteoarthritic knees with unicompartmental arthritis. J Bone Joint Surg Br. 1998 Sep;80(5):862-5. doi: 10.1302/0301-620x.80b5.8835. PMID 9768899
- [Background] NAR. The Norwegian Arthroplasty Register. 2013.
- [Background] NZJR. The New Zealand Joint Registry. Fifteen year report January 1999 to December 2013. 2014.
- [Background] Pandit H, Liddle AD, Kendrick BJ, Jenkins C, Price AJ, Gill HS, Dodd CA, Murray DW. Improved fixation in cementless unicompartmental knee replacement: five-year results of a randomized controlled trial. J Bone Joint Surg Am. 2013 Aug 7;95(15):1365-72. doi: 10.2106/JBJS.L.01005. PMID 23925740
- [Background] Liddle AD, Pandit H, O'Brien S, Doran E, Penny ID, Hooper GJ, Burn PJ, Dodd CA, Beverland DE, Maxwell AR, Murray DW. Cementless fixation in Oxford unicompartmental knee replacement: a multicentre study of 1000 knees. Bone Joint J. 2013 Feb;95-B(2):181-7. doi: 10.1302/0301-620X.95B2.30411. PMID 23365026
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417
- [Background] Collins NJ, Roos EM. Patient-reported outcomes for total hip and knee arthroplasty: commonly used instruments and attributes of a "good" measure. Clin Geriatr Med. 2012 Aug;28(3):367-94. doi: 10.1016/j.cger.2012.05.007. Epub 2012 Jun 22. PMID 22840304
- [Background] Beard DJ, Harris K, Dawson J, Doll H, Murray DW, Carr AJ, Price AJ. Meaningful changes for the Oxford hip and knee scores after joint replacement surgery. J Clin Epidemiol. 2015 Jan;68(1):73-9. doi: 10.1016/j.jclinepi.2014.08.009. Epub 2014 Oct 31. PMID 25441700
- [Background] Andersen LO, Husted H, Otte KS, Kristensen BB, Kehlet H. High-volume infiltration analgesia in total knee arthroplasty: a randomized, double-blind, placebo-controlled trial. Acta Anaesthesiol Scand. 2008 Nov;52(10):1331-5. doi: 10.1111/j.1399-6576.2008.01777.x. PMID 19025523
- [Background] Kerr DR, Kohan L. Local infiltration analgesia: a technique for the control of acute postoperative pain following knee and hip surgery: a case study of 325 patients. Acta Orthop. 2008 Apr;79(2):174-83. doi: 10.1080/17453670710014950. PMID 18484242
- [Derived] Knifsund J, Niinimaki T, Nurmi H, Toom A, Keemu H, Laaksonen I, Seppanen M, Liukas A, Pamilo K, Vahlberg T, Aarimaa V, Makela KT. Functional results of total-knee arthroplasty versus medial unicompartmental arthroplasty: two-year results of a randomised, assessor-blinded multicentre trial. BMJ Open. 2021 Jun 23;11(6):e046731. doi: 10.1136/bmjopen-2020-046731. PMID 34162649